CLINICAL TRIAL: NCT06615713
Title: A Prospective Study to Evaluate the Safety and Effectiveness of Steerable Ureteroscopic Renal Evacuation (SURE) Using the CVAC® Set
Brief Title: Evaluate the Safety and Effectiveness of Steerable Ureteroscopic Renal Evacuation (SURE) Using the CVAC® System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Calyxo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP00003
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Renal Stones; Kidney Stone; Urolithiasis
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi; Urolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Steerable Ureteroscopic Renal Evacuation (SURE) with CVAC System (Experimental): The CVAC Aspiration System is a sterile, single use, steerable ureteral catheter system with integrated vision, irrigation and aspiration for the treatment and removal of urinary stones (kidney stones, fragments, and dust).
  Interventions: Device: Steerable Ureteroscopic Renal Evacuation (SURE) with CVAC System

INTERVENTIONS:
Device: Steerable Ureteroscopic Renal Evacuation (SURE) with CVAC System — The CVAC Aspiration System is a sterile, single use, steerable ureteral catheter system with integrated vision, irrigation and aspiration for the treatment and removal of urinary stones (kidney stones, fragments, and dust).

SUMMARY:
The purpose of the study is to assess safety and efficacy of a novel steerable ureteral catheter system, the CVAC System for the treatment of urinary stones.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for ureteroscopy with laser lithotripsy;
* Be willing and able to return for and respond to all study-related follow up procedures; and,
* Have been informed of the nature of the study and have agreed to the IRB approved informed consent form (ICF).

Exclusion Criteria:

* Significant morbidities;
* Unable to meet the treatment and follow up protocol requirements; and,
* Ureteral or kidney abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Stone Clearance | Day 1 and Day 30
  The stone clearance at Post-Op Day 1 (POD1) and Post-Op Day 30 (POD30) on non-contrast CT (NCCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Muljibhai Patel Urological Hospital, Nadiād, India